CLINICAL TRIAL: NCT07031739
Title: Sequential Multiple Assignment Randomized Trial to Reduce Food Insecurity and Improve Adherence in Patients With Hypertension
Brief Title: Sequential Multiple Assignment Randomized Trial to Reduce Food Insecurity
Acronym: SMART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB00115742; 1R01HL173064-01A1 (NIH)
Record Dates: First submitted 2025-06-05; First posted 2025-06-22 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-05

CONDITIONS: Uncontrolled Hypertension
Keywords: cardiovascular disease; hypertension; Food insecurity
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension | interventions — Community Health Workers; Insemination, Artificial, Heterologous

STUDY DESIGN:
Intervention Model Description: Assignment Randomized Trial to reduce Food Insecurity and Improve Adherence in Patients with Hypertension (SMART-FI) is a single-site, open-label, longitudinal two-stage SMART. Participants will be randomized to one of two first-stage treatments for 3 months: 1) information about community resources or 2) in-person community health workers (CHW) support. Participants who do not have a 10mmHg improvement in systolic blood pressure (SBP) at 3 months will be re-randomized to one of two second-stage treatments for an additional 3 months: 1) CHW support or 2) home delivery of medically tailored meals (MTM).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Resource information (Experimental): Participants randomized to this arm will receive a tailored list of information about community resources. The list will include information about local food resources (e.g. local food pantries) and government programs (e.g. Supplemental Nutrition Assistance Program) to address Food Insecurities (FI).
  Interventions: Behavioral: Resource information
- Community Health Worker (CHW) assistance (Experimental): The CHW will meet with the participant at the baseline visit and will follow up with participants at least every other week. The CHW will also work directly with the patient's care team. As health advisors, CHW will help them overcome commonly experienced barriers in blood pressure management.
  Interventions: Behavioral: Community Health Worker (CHW) assistance
- Medically-tailored Meals (MTM) (Experimental): MTM will consist of weekly home meal delivery. During the 3 months, participants will receive 10 medically tailored refrigerated or frozen meals (5 lunches and 5 dinners) delivered to their home weekly. All meals are planned by a registered dietician and based on the Dietary Approaches to Stop Hypertension (DASH) diet.
  Interventions: Behavioral: Medically-tailored Meals (MTM)

INTERVENTIONS:
Behavioral: Resource information — Participants randomized to this arm will receive a tailored list of information about community resources.
  Other Names: information about local food resources
  Arms: Resource information
Behavioral: Community Health Worker (CHW) assistance — The CHW will meet with the participant at the baseline visit and will follow up with participants at least every other week. The CHW will also work directly with the patient's care team.
  Other Names: community advocates
  Arms: Community Health Worker (CHW) assistance
Behavioral: Medically-tailored Meals (MTM) — MTM will consist of weekly home meal delivery. During the 3 months, participants will receive 10 medically tailored refrigerated or frozen meals (5 lunches and 5 dinners) delivered to their home weekly.
  Other Names: meals are planned by a registered dietician
  Arms: Medically-tailored Meals (MTM)

SUMMARY:
Food insecurity affects 20% of the 116 million people in the US with hypertension and is associated with poor adherence to evidence-based treatments and disparities in hypertension outcomes. Interventions are being used to address food insecurity in clinical care settings, but people differ in the support they need to reduce food insecurity and little is known about which food insecurity interventions work best, or for whom. The goal of this study is to develop and test an adaptive food insecurity intervention using a Sequential Multiple Assignment Randomized Trial to determine which initial food insecurity intervention is more effective in improving adherence and blood pressure in patients with hypertension and for those who do not respond to the initial intervention, evaluate how to best provide additional support.

DETAILED DESCRIPTION:
In the US, 47% of adults have hypertension (HTN), and HTN is the leading cause of cardiovascular disease morbidity and mortality. Uncontrolled HTN increases the risk of cardiovascular disease, chronic kidney disease, and cognitive impairment. Current guidelines recommend the adoption of a healthy diet as an integral part of ongoing treatment regardless of the underlying antihypertensive drug treatment. The Dietary Approaches to Stop Hypertension (DASH) eating pattern is a diet rich in fruits, vegetables, and whole grains with a reduced content of sodium and saturated fat. The DASH is the diet with the strongest evidence to be effective for lowering blood pressure. Despite the evidence base for the effectiveness of DASH as well as pharmacological treatments, economic factors are common barriers to individuals with HTN adhering to treatments. Adherence is multidimensional and involves initiation, implementation, and persistence. Food insecurity (FI), the lack of consistent access to the food needed for a healthy life, is an important factor that leads to HTN disparities. Individuals living in food insecure households are less likely to adhere to prescribed HTN treatments, such as DASH and medications, and more likely to have worse blood pressure control.

Because of the prevalence of FI and associated poor health outcomes, a growing number of health systems and health insurers are investing in integrating interventions to address FI as part of routine clinical care. These interventions include 1) providing information to patients about community resources), 2) utilizing community health workers (CHW), and 3) home delivery of medically tailored meals (MTM). Studies have shown these FI interventions have varying levels of success on improving food security and health. However, people often need varying levels of support to address needs, and, rather than using only one single intervention to address FI, there remains a gap in understanding whether adaptively allocating resources based on need has the potential to more effectively, equitably, and efficiently improve food security and health for a greater proportion of patients.

To advance the science in patient adherence and blood pressure management, this study will conduct a sequential multiple assignment randomized trial (SMART) among food-insecure patients with uncontrolled HTN. SMART uses experimental design principles to determine whether and how to alter treatments to build optimal adaptive interventions. This study will assess the change in adherence and blood pressure over time (0-9 months). This study will also evaluate if treatment options were more effective for particular patients. Several other measures are included in this study to learn more about how an adaptive intervention designed to address FI affects blood pressure, adherence, food security, health-related quality of life, and other key risk factors for blood pressure control in patients with HTN.

The proposed Sequential Multiple Assignment Randomized Trial to reduce Food Insecurity and Improve Adherence in Patients with Hypertension (SMART-FI) is a single-site, open-label, longitudinal two-stage SMART. Participants will be randomized to one of two first-stage treatments for 3 months: 1) information about community resources or 2) in-person CHW support. Participants who do not have a 10mmHg improvement in systolic blood pressure (SBP) at 3 months will be re-randomized to one of two second-stage treatments for an additional 3 months: 1) CHW support or 2) home delivery of MTM. The study will recruit 224 participants for this trial. Participants will engage in the interventions up to 6 months and will be followed for a total of 9 months. In Aim 1, the study will determine which first-stage FI intervention is more effective in improving adherence and blood pressure. In Aim 2, the study will evaluate which FI intervention is the best next step for those who do not respond to the initial intervention. In Aim 3, the study will explore how, why, and under what circumstances participants achieved improvements to the first- and second-stage interventions by conducting semi-structured interviews with participants and evaluating for potential predictors of heterogeneity in response to each intervention.

ELIGIBILITY:
Inclusion Criteria:

* Must Speak English or Spanish
* have a diagnosis of Hypertension (HTN)
* prescribed at least one blood pressure lowering medication (including thiazide diuretic, calcium channel blocker, beta-blocker, angiotensin-converting enzyme inhibitors, or angiotensin receptor blocker)
* past 2 blood pressures at their primary care doctor were greater than or equal to130/80mmHg (millimeters of Mercury)
* seen by their primary care doctor in the past 6 months
* experience Food Insecurities (FI) based on the 2-item Hunger Vital Sign

Exclusion Criteria:

* Systolic Blood Pressure > 210mmHg or a diastolic blood pressure > 120mmHg
* have a severe cognitive impairment or major psychiatric illness that prevents consent or serious medical condition which either limits life expectancy or requires active management (e.g. certain cancers)
* pregnant, breastfeeding, or planning to become pregnant in the next 6 months
* planning on moving out of the area within 6 months
* lack safe stable housing
* do not have the ability to store meals
* lack of a telephone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Systolic blood pressure value | Month 9
  Systolic blood pressure measured as mmHg
Diastolic blood pressure value | Month 9
  Diastolic blood pressure measured as mmHg
Dietary Approaches to Stop Hypertension (DASH) diet adherence Score | Month 9
  Change in DASH diet adherence over time, based on the Mellen DASH diet adherence index - The Mellen DASH diet index is a nutrient-based method for assessing adherence to the Dietary Approaches to Stop Hypertension (DASH) diet. It uses nine key nutrients to determine a score ranging from 0 to 9, with 9 indicating the most adherence - Food items on the FFQ are assigned to 7 DASH food groups and 3 components using the Harvard nutrient database. Servings in each component are scored 0, 0.5, and 1. The DASH diet adherence score ranges from 0 to 10 and is the sum of the 10 component scores. Higher scores indicate greater diet concordance.
Medication adherence Score | Month 9
  Change in medication adherence based on the 12-item Adherence to Refills and Medications Scale - The 12-item Adherence to Refills and Medications Scale (ARMS) is a self-report questionnaire designed to measure a patient's adherence to medication regimens - Each scale comprises five items that are scored on a Likert-type scale, where 1 = strongly disagree, 2 = disagree, 3 = uncertain, 4 = agree and 5 = strongly agree. Higher scores indicate stronger beliefs in the necessity of medication and greater concerns about taking it.
Food Security Score | Month 9
  Change in food security over time based on the 10-item USDA Food Security Survey Module with a 30-day reference period - The USDA Food Security Survey Module (HFSSM) uses a 10-item adult-referenced module to assess food security status. A raw score is calculated based on affirmative responses to these 10 questions, and this score is then used to classify households into food security categories: high, marginal, low, or very low.
  High Food Security (Raw Score 0): No affirmative responses. Marginal Food Security (Raw Score 1-2): One or two affirmative responses. Low Food Security (Raw Score 3-5): Three to five affirmative responses. Very Low Food Security (Raw Score 6-10): Six to ten affirmative responses.

SECONDARY OUTCOMES:
Health-related quality of life Score | Month 9
  Change in EQ-5D-5L scores - assigning a numerical value to each response level (i.e., 1 for "no problems", 5 for "extreme problems"/"unable to") and summing these values across the five items, resulting in a score from 5 (11,111, no problems on any dimension) to 25 (55,555, extreme problems on all dimensions)
Number of Changes in Community resource Use | Month 9
  Changes in use of community resources (e.g. food pantries, supplemental nutrition assistance program)

OTHER OUTCOMES:
Change in Food expenditure Amount | Month 9
  Out-of-pocket monthly food expenditures
Adherence Rate to medically tailored meal consumption (MTM) | Month 3
  Food consumption diaries -Adherence to medically tailored meals
Change in Depressive symptoms Score | Month 9
  Change in depressive symptoms based on the Patient Health Questionnaire-8 (PHQ-8) over time - PHQ-8 Scoring The Patient Health Questionnaire-8 (PHQ-8) is a screening tool used to assess the severity of depressive symptoms.
  Scoring Instructions:
  Each question is rated on a scale of 0 (not at all) to 3 (nearly every day). Add up the scores for all 8 questions. The total score ranges from 0 to 24.
  Interpretation:
  0-4: No significant symptoms of depression. 5-9: Mild depression. 10-14: Moderate depression. 15-19: Moderately severe depression. 20-24: Severe depression.
Change in Stress Score | Month 9
  Change in stress based on the Change in stress based on the Perceived Stress Scale scores - The Perceived Stress Scale (PSS) score provides insights into an individual's perceived stress levels. Higher scores generally indicate greater perceived stress, while lower scores suggest lower stress. The PSS-10, a shortened version of the PSS, ranges from 0 to 40, with scores typically categorized as low (0-13), moderate (14-26), and high (27-40) stress.
Change in Hypertension (HTN) management Score | Month 9
  Change in scores in hypertension self-management behaviors based on the HTN self-care profile - The Hypertension Self-Care Profile (HBP SCP) is a questionnaire used to assess an individual's self-care behaviors related to managing hypertension. It's a multi-scale instrument, meaning it includes different sections to assess different aspects of self-care, including behavior, motivation, and self-efficacy - A high score on the HBP SCP generally indicates that an individual is actively engaged in self-care behaviors that are important for managing hypertension, has a strong motivation to engage in these behaviors, and has a high degree of confidence in their ability to manage their condition.
Change in Number of Healthcare uses | Months 3, 6, and 9
  The measure will assess differences in the number of missed appointments, emergency department use, and hospitalizations from baseline to follow at 3, 6 and 9 months. The study will assess differences in the number of missed appointments and visits between the arms

CONTACTS AND LOCATIONS:
Overall Officials: Deepak Palakshappa, MD, MSHP, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No